CLINICAL TRIAL: NCT02841865
Title: Evaluation of Radiological Response of Pancreatic Neuroendocrine Tumors: Comparison Between the Choi and the RECIST Criteria
Brief Title: Radiological Response of Pancreatic Neuroendocrine Tumors: Comparison Between the Choi and the RECIST Criteria
Acronym: CRIPNET
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Other Study IDs: GET-SUN-2015-01
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The Response Evaluation Criteria in Solid Tumors (RECIST), based on differences in tumor size, has been considered as a reproducible method that facilitates not only the measurement of the mass but the evaluation of response to given treatments; while classic chemotherapy induces a reduction of the tumor, new target therapies frequently produce the stabilization of the disease or a delayed progression. These new therapeutic alternatives have shade light on the limitations of the RECIST criteria, since the response to these type of treatments are basically associated with changes on the radiological characteristics of the tumor, as well as other findings in functional imaging.

This study is aimed to compare the response rates according both Choi and RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pancreatic neuroendocrine tumor with a Ki67 index <20%, who accept to participate and sign the consent form. In case of death patients, waiver of consent has been considered.
* Patients who, according daily clinical practice, have been treated with sunitinib between February 2012 to end of inclusion period, with a follow up of at least 6 months.
* Patients with a baseline imaging study (TC with arterial phase) and, at least, a 6-months follow-up evaluation. Patients with progression or exitus before the first imaging evaluation will not be included.

Exclusion Criteria:

* Patients with a follow-up of <6months because of any other cause beyond progression of disease or exitus.
* Patients without a baseline radiological evaluation or at 3/6 months.
* Patients who do not accept to participate in the study.
* Patients with anti-angiogenic treatment within 3 months prior to the start of sunitinib treatment.
* Patients treated with sunitinib plus any other anti-proliferative agent beyond ASS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a neuroendocrine pancreatic tumor, treated with sunitinib, with at least one radiological evaluation every 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 3 months
  According Choi and RECIST Criteria

SECONDARY OUTCOMES:
Progression Free Survival on partial response | 3 months
  Time between start of treatment and progression of disease in patients with partial response
Progression Free Survival on Stable Disease | 3 months
  Time between start of treatment and progression of disease in patients with stable disease
Impact of Tumor Uptake on Response to Treatment | 3 months
  Description of the uptake of pancreatic neuroendocrine tumor lesions in the arterial phase (baseline evaluation), and assessment of a possible correlation with the response to treatment using the RECIST criteria.
Impact of Response to Treatment and Progression Free Survival | 3 months
  Description of the uptake of pancreatic neuroendocrine tumor lesions in the arterial phase and assess ment of a possible correlation with the progression free survival.
Impact of Choi criteria and Progression of Disease | 3 months
  Correlation of Changes on the uptake of pancreatic neuroendocrine tumor lesions in the arterial phase and progression of disease.

CONTACTS AND LOCATIONS:
Overall Officials: María del Pilar Solís Hernández, M.D., Study Chair — Hospital Universitario Central de Asturias; Paula Jiménez Fonseca, M.D., Study Chair — Hospital Universitario Central de Asturias; David Calvo Temprano, M.D., Study Chair — Hospital Universitario Central de Asturias
Locations (10):
- Spain (10):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No